CLINICAL TRIAL: NCT02814227
Title: Wireless Sensor Patch for Reducing Barriers to In-home Sleep Apnea Screening
Brief Title: Validation of Sleep Apnea Screening Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Zansors (Industry)
Responsible Party: Principal Investigator, J. Todd Arnedt, Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R41MD008845-01 (NIH)
Record Dates: First submitted 2015-10-25; First posted 2016-06-27 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea screening device
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zansors® sleep screening device (Experimental): Zansors device compared to overnight polysomnography
  Interventions: Device: Zansors® sleep screening device

INTERVENTIONS:
Device: Zansors® sleep screening device — Intervention is the validation of a sleep apnea screening device against the gold-standard assessment of in-laboratory polysomnography

SUMMARY:
Obstructive sleep apnea (OSA) is the most common type of sleep apnea. OSA affects an estimated 18-40 million adults and 0.7-3% of all children in the US. The marketplace currently does not have an affordable, easy-to-use, over-the-counter, home-based OSA screening device. An affordable, available, FDA-approved and easy-to-use over-the-counter OSA screening tool would allow greater screening of at-risk individuals, especially in underserved communities with low socioeconomic status, hopefully encouraging a greater proportion of such individuals to seek treatment for their condition. The specific goal of this project is to compare the Zansors® micro sleep sensor screening device against gold-standard polysomnography to establish the device's preliminary validity to screen for OSA accurately.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) results in tiredness, depression and fatigue, and has several associated common comorbidities. It is believed that over 80% of OSA remains undiagnosed. Poorer and disadvantaged communities are at higher risk for sleep disorders, including OSA, even after accounting for other risk factors. The gold-standard method for diagnosing OSA is in-laboratory polysomnography; however, this procedure is generally available only to patients with health insurance due to its high cost. As a result, communities at particularly high risk for OSA are less likely to have this serious sleep disorder appropriately diagnosed and treated.

An affordable, available, FDA-approved and easy-to-use over-the-counter OSA screening tool would allow greater screening of at-risk individuals, especially in underserved communities with low socioeconomic status, hopefully encouraging a greater proportion of such individuals to seek treatment for their condition. Zansors® has developed a bioengineered, semiconductor prototype that measures breathing and movement during sleep. It is a 1.5 x 2.5 x 0.2 inch wireless package using four key technologies:

1. an adjustable microphone;
2. a 3-axis accelerometer;
3. embedded algorithms to measure sleep events; and
4. acrylic adhesive.

The product will be designed as an FDA-approved over-the-counter device that the patient can wear during sleep and wake up with a color score of red, yellow, or green depending on their sleep apnea status. The features of this product include that it is home-based; easy to use; non-invasive; wireless; disposable; low cost ($20-50); and presents easily understandable test results. However, such a device must first be validated against gold-standard polysomnography.

The specific goal of this project is to compare the Zansors® micro sleep sensor screening device against gold-standard polysomnography to establish the device's preliminary validity to screen for OSA accurately.

ELIGIBILITY:
Inclusion Criteria:

* Must be over 18 and referred by medical staff for an overnight assessment for suspected sleep apnea

Exclusion Criteria:

* Pregnancy
* Heart disease including congestive heart failure or a pacemaker
* Breathing disorder (emphysema or chronic obstructive breathing disorder)
* Neurological disorder such as Parkinson's Disease
* Restless leg syndrome or Periodic limb movement
* Allergies to metal
* Pre-existing skin conditions where sensor would be attached

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Todd Arnedt, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zansors® Sleep Screening Device
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Zansors® Sleep Screening Device
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Specificity
Description: Specificity of Zansors' device to detect apnea events compared to gold-standard polysomnography over an 8-hour period of sleep at 30-second intervals
Time Frame: 8 hours
Measure: Number; unit: percentage of true negatives
Arm/Group | Zansors® Sleep Screening Device
Number analyzed (Participants) | 52
percentage of true negatives | 71.4

2. Secondary Outcome: Sensitivity
Description: Sensitivity of Zansors' device to detect apnea events compared to gold-standard polysomnography over an 8-hour period of sleep at 30-second intervals
Time Frame: 8 hours
Measure: Number; unit: percentage of true positives
Arm/Group | Zansors® Sleep Screening Device
Number analyzed (Participants) | 52
percentage of true positives | 75

3. Secondary Outcome: Positive Predictive Value (PPV)
Description: PPV of Zansors' device to detect apnea events compared to gold-standard polysomnography over an 8-hour period of sleep at 30-second intervals
Time Frame: 8 hours
Measure: Number; unit: positive predictive value
Arm/Group | Zansors® Sleep Screening Device
Number analyzed (Participants) | 52
positive predictive value | 0.692

4. Secondary Outcome: Negative Predictive Value (NPV)
Description: NPV of Zansors' device to detect apnea events compared to gold-standard polysomnography over an 8-hour period of sleep at 30-second intervals
Time Frame: 8 hours
Measure: Number; unit: negative predictive value
Arm/Group | Zansors® Sleep Screening Device
Number analyzed (Participants) | 52
negative predictive value | 0.77

ADVERSE EVENTS:
Time Frame: 8 hours
Arm/Group | Zansors® Sleep Screening Device
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes